CLINICAL TRIAL: NCT00549809
Title: Comparison Between IMV and SIMV/PS for Ventilatory Support of Children: a Randomized Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: José Roberto Fioretto, UNESP - Botucatu Medical School
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-04
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Respiratory Failure
Keywords: mechanical ventilation; respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMV, SIMV (Active Comparator)
  Interventions: Procedure: Intermittent mandatory ventilation (IMV) and synchronous IMV

INTERVENTIONS:
Procedure: Intermittent mandatory ventilation (IMV) and synchronous IMV — Patients divided to receive two different modes of mechanical ventilation.
  Other Names: IMV (intermittent mandatory ventilation); SIMV (synchronous intermittent mandatory ventilation)

SUMMARY:
Objectives: to compare intermittent mandatory ventilation (IMV) with synchronous intermittent mandatory ventilation associated with pressure support (SIMV/PS) related to duration of mechanical ventilation/weaning and length of stay in PICU (LS). Design: randomized clinical trial. Setting: Pediatric intensive care unit at a university-affiliated hospital.

DETAILED DESCRIPTION:
Objectives: to compare intermittent mandatory ventilation (IMV) with synchronous intermittent mandatory ventilation associated with pressure support (SIMV/PS) related to duration of mechanical ventilation/weaning and length of stay in PICU (LS). Design: randomized clinical trial. Setting: Pediatric intensive care unit at a university-affiliated hospital. Patients: children between 28 days and 4 years old, admitted between 10/2002 and 06/2004, and receiving mechanical ventilation (MV) for more than 48 hours. Patients were randomly assigned into two groups: IMV (IMVG; n=35) and SIMV/PS (SIMVG; n=35). Children with acute respiratory distress syndrome and tracheostomy were excluded. Ventilation and oxygenation data were recorded at admission and beginning of weaning. Results: Groups were not statistically different for age, gender, MV indications, PRISM score, COMFORT scale, sedatives, and ventilation and oxygenation parameters. Median of MV duration was 5 days for both groups (p>0.05). Also, there were no statistical differences for duration of weaning [IMVG: 1 day (1 - 6) vs. SIMVG: 1 day (1 - 6); p>0.05] and LS [IMVG: 8 days (2 - 22) vs. SIMVG: 6 days (3 - 20); p>0.05]. Conclusion: There was no statistically significant difference between IMV and SIMV/PS in these children related to MV and weaning duration, and PICU length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 28 days and four years, who were consecutively admitted to the PICU and required MV for more than 48h were included.

Exclusion Criteria:

* Children who had chronic respiratory failure, tracheostomy, those transferred from the hospital, or died were excluded as were patients with acute respiratory distress syndrome (ARDS).

Ages: 28 Days to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2005-10; Primary Completion 2007-02 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
duration of mechanical ventilation/weaning and length of stay in PICU | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Fioretto, MD, PhD, Principal Investigator — UNESP - Botucatu Medical School
Locations (1):
- Jose Roberto Fioretto, Botucatu, São Paulo, Brazil

REFERENCES:
- [Derived] Moraes MA, Bonatto RC, Carpi MF, Ricchetti SM, Padovani CR, Fioretto JR. Comparison between intermittent mandatory ventilation and synchronized intermittent mandatory ventilation with pressure support in children. J Pediatr (Rio J). 2009 Jan-Feb;85(1):15-20. doi: 10.2223/JPED.1849. Epub 2008 Nov 6. English, Portuguese. PMID 18989547